CLINICAL TRIAL: NCT05296733
Title: A Non-randomised, Open-label, 2-part, Parallel-cohort Trial to Evaluate 1) Pharmacokinetics, Safety, and Tolerability of a Single Subcutaneous Dose of BI 456906 in Patients With Cirrhosis and Varying Degrees of Hepatic Impairment Relative to Healthy Subjects With and Without Overweight/Obesity and 2) Safety and Tolerability of Multiple Subcutaneous Doses of BI 456906 in Patients With Overweight/Obesity With Cirrhosis and Varying Degrees of Hepatic Impairment Relative to Patients With Overweight/Obesity Without Cirrhosis/Hepatic Impairment
Brief Title: A Study to (1) Compare How BI 456906 is Taken up in the Body of Healthy People and People With Liver Problems and (2) Find Out How People With Overweight and Obesity, With and Without Liver Problems, Tolerate Different Doses of BI 456906
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1404-0010; 2021-006247-10 (EudraCT Number)
Record Dates: First submitted 2022-03-23; First posted 2022-03-25 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Healthy; Liver Diseases; Obesity
MeSH Terms: conditions — Liver Diseases; Obesity | interventions — BI 456906

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part A: BI 456906: Cohort 1 (Experimental): Healthy subjects
  Interventions: Drug: BI 456906
- Part A: BI 456906: Cohort 2 (Experimental): Patients with cirrhosis + Child-Turcotte-Pugh (CTP) Class A
  Interventions: Drug: BI 456906
- Part A: BI 456906: Cohort 3 (Experimental): Patients with cirrhosis + CTP Class B
  Interventions: Drug: BI 456906
- Part A: BI 456906: Cohort 4 (Experimental): Patients with cirrhosis + CTP Class C
  Interventions: Drug: BI 456906
- Part B: BI456906: Cohort 1 (Experimental): Patients with overweight/obesity without cirrhosis/hepatic impairment
  Interventions: Drug: BI 456906
- Part B: BI456906: Cohort 2 (Experimental): Patients with overweight/obesity with cirrhosis + CTP Class A
  Interventions: Drug: BI 456906
- Part B: BI456906: Cohort 3 (Experimental): Patients with overweight/obesity with cirrhosis + CTP Class B
  Interventions: Drug: BI 456906

INTERVENTIONS:
Drug: BI 456906 — BI 456906
  Other Names: survodutide

SUMMARY:
This study is open to adults who have different levels of liver problems and adults who are healthy. People with or without overweight or obesity can take part.

This study has 2 parts. The purpose of Part 1 is to find out whether having liver problems influences how BI 456906 is taken up in the body. The purpose of Part 2 is to find out whether having liver problems influences how people with overweight and obesity tolerate different doses of BI 456906.

In Part 1, participants get a single injection of BI 456906 under their skin and stay at the study site for 2 nights afterwards. They are in the study for about a month. During this time, they visit the study site about 8 more times. The doctors compare the amount of BI 456906 in the blood of healthy people and people with liver problems.

In Part 2, participants get 1 or 2 injections of BI 456906 once a week under their skin for 28 weeks. At the beginning, they get lower doses of BI 456906. Over time, they get higher doses until they reach a certain dose of BI 456906. This dose is then maintained until the end of the treatment. Participants in Part 2 are in the study for about 7 months. During this time, they visit the study site about 16 times and get about 15 phone calls from the site staff. The doctors record the number of people with health problems that could have been caused by treatment with BI 456906. They compare the results between participants with liver problems and those without liver problems.

In both parts, doctors also regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion Criteria -Part A:

* Male or female subjects with age ≥18 years (or the minimum country specific age of consent if >18 years) and 75 years, inclusive at the screening visit.
* Body mass index (BMI) of 18.5-40.0 kg/m2 (inclusive).
* Signed and dated written informed consent in accordance with International Council on Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial.
* Women of childbearing potential must be willing and able to use two forms of effective contraception where at least one form is highly effective method of birth control per ICH M3 (R2) that results in a low failure rate (i.e. <1% per year when used consistently and correctly). A list of contraception methods meeting these criteria is provided in the subject information. Please note that oral contraceptives are not allowed during the treatment period.

A woman is considered of childbearing potential, i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. Tubal ligation is NOT a method of permanent sterilisation. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause.

Further inclusion criteria apply.

-Part B:

* Male or female subjects between the ages of ≥18 (or the minimum country specific age of consent if >18 years) and 75 years, inclusive, at the screening visit.
* Subjects with overweight or obesity, defined as BMI ≥27 kg/m2 at the screening visit.
* A minimum absolute body weight of 70 kg for females and 80 kg for males at the screening visit.
* Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial.

Further inclusion criteria apply.

Exclusion criteria -Part A:

* Estimated Glomerular Filtration Rate (eGFR) <60 mL/min/1.73 m2 (Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] formula).
* Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome type 2, manifest hypo- or hyperthyroidism at screening.
* Calcitonin ≥20 pg/mL (5.84 pmol/L) at the screening visit.
* History of chronic or acute pancreatitis or elevation of serum lipase/amylase >2×ULN, or fasting serum triglyceride levels of >500 mg/dL (>5.65 mmol/L) at screening.

Further exclusion criteria apply.

-Part B:

* Prior surgery of the gastrointestinal tract that could interfere with body weight (including minimally invasive/endoscopic bariatric devices, bariatric surgery including metabolic operation that involves resection and/or reconstruction of any portion of the gastrointestinal tract) except appendectomy and simple hernia repair before randomization. However, a subject previously treated with reversible weight loss devices such as gastric banding, or intragastric balloon and removed longer than 12 months before screening should not be excluded.
* Glycosylated Hemoglobin, Type A1 (HbA1c) ≥11% at screening or diagnosed with type 1 diabetes mellitus.
* Exposure to Glucagon-like-peptide 1 (GLP-1) receptor agonist-based therapies (within 3 months prior to screening or within 5 half-lives of the drug, whichever is longer).
* Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome type 2, manifest hypo- or hyperthyroidism at screening.

Further exclusion criteria apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2022-04-27 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2023-12-29 (Actual)

PRIMARY OUTCOMES:
Part A: Area under the concentration-time curve of BI 456906 in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | Up to 360 hours
Part A: Maximum measured concentration of BI 456906 in plasma (Cmax) | Up to 360 hours
Part B: Percentage of patients treated who experience treatment-emergent adverse event | Up to Day 218

SECONDARY OUTCOMES:
Part A: Percentage of patients treated who experience treatment-emergent adverse event | Up to Day 35

CONTACTS AND LOCATIONS:
Locations (13):
- United States (5):
  - Arizona Liver Health, Chandler, Arizona
  - Covenant Metabolic Specialists, LLC, Fort Myers, Florida
  - Covenant Metabolic Specialists, LLC, Sarasota, Florida
  - American Research Corporation at the Texas Liver Institute, San Antonio, Texas
  - IMA Clinical Research San Antonio, San Antonio, Texas
- Germany (3):
  - Universitätsklinikum Bonn AöR, Bonn
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum Ulm, Ulm
- Hungary (2):
  - Semmelweis University, Budapest
  - CRU Hungary Ltd., Kistarcsa
- New Zealand Clinical Research (NZCR), Auckland, New Zealand
- Dr. Piotr Napora, Center of Clinical Research, Wroclaw, Poland
- SUMMIT CLINICAL RESEARCH, s.r.o., Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- [Derived] Lawitz EJ, Fraessdorf M, Neff GW, Schattenberg JM, Noureddin M, Alkhouri N, Schmid B, Andrews CP, Takacs I, Hussain SA, Fenske WK, Gane EJ, Hosseini-Tabatabaei A, Sanyal AJ, Mazo DF, Younes R; NCT05296733 Investigators. Efficacy, tolerability and pharmacokinetics of survodutide, a glucagon/glucagon-like peptide-1 receptor dual agonist, in cirrhosis. J Hepatol. 2024 Nov;81(5):837-846. doi: 10.1016/j.jhep.2024.06.003. Epub 2024 Jun 8. PMID 38857788
- See also: Related Info — https://www.mystudywindow.com/